CLINICAL TRIAL: NCT01834300
Title: The Effects of Exercise Training on Visceral Fat, Insulin Sensitivity, Β-cell Function and Triglyceride Kinetics in Patients with Non-alcoholic Fatty Liver Disease (NAFLD).
Brief Title: The Effect of Exercise Intervention on Insulin Resistance in Non-alcoholic Fatty Liver Disease (NAFLD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: Royal Liverpool University Hospital (Other Government); University of Surrey (Other); Imperial College London (Other); Royal Surrey County Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09/H1008/1
Record Dates: First submitted 2013-04-12; First posted 2013-04-17 (Estimated); Last update posted 2024-12-18 (Actual); Status verified 2024-05

CONDITIONS: Non Alcoholic Fatty Liver Disease
Keywords: Hepatic insulin sensitivity; Muscle insulin sensitivity; B cell function; VLDL1 TG metabolism; VLDL2 TG metabolism
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Experimental): Unsupervised exercise training This group will be given 1 hour lifestyle counseling by the exercise trainer after which they will have no contact with the exercise trainer to the end of the intervention period. The exercise intervention will be offered to the subjects once the post studies are completed.
  Interventions: Behavioral: Unsupervised exercise training
- lifestyle counseling and exercise (Experimental): Supervised exercise training Four months exercise training intervention will be either gym-based or patients will choose the mode of exercise that suits their lifestyle. Patients will be encouraged to exercise four times per week for 30-45 min at 60-80 % of maximal heart rate, with a 5 min warm-up and warm-down. Participants will be given free access to a variety of affiliated sports centres and will use the Wellness Key system, a software program that enables researchers to remotely track the exercise activity of participants very accurately. To ensure compliance with rest or exercise, all participants of both groups will have their mean physical activity level in 2 non-consecutive weeks evaluated with an ambulatory accelerometer.
  Interventions: Behavioral: Supervised exercise training

INTERVENTIONS:
Behavioral: Unsupervised exercise training — The patients will be given lecture on lifestyle changes and its benefitial effects on health at the begining of the study by the exercise trainer. There will be no conatct with the exercise trainer for the period of intervention for 4 months.
  Arms: Control
Behavioral: Supervised exercise training — Patients will be encouraged to exercise four times per week for 30-45 min at 60-80 % of maximal heart rate, with a 5 min warm-up and warm-down. Participants will be given free access to a variety of affiliated sports centres and will use the Wellness Key system, a software program that enables researchers to remotely track the exercise activity of participants very accurately. To ensure compliance with rest or exercise, all participants of both groups will have their mean physical activity level in 2 non-consecutive weeks evaluated with an ambulatory accelerometer.
  Arms: lifestyle counseling and exercise

SUMMARY:
This project examines the effects of a 4 month structured exercise intervention program in patients with non-alcoholic fatty liver disease (NAFLD). We will examine changes in total and depot-specific (i.e.in different tissues, liver, muscle and pancreas)fat. We will correlate these with measurements of the insulin from the liver. The hypothesis is that by reducing fat in these specific depots we can reduce insulin resistance and prevent progression to diabetes.

DETAILED DESCRIPTION:
1. Exercise program: We are asking people to take part in a supervised exercise program for 4 months. This involves on average a weekly supervised exercise bout plus other unsupervised exercise bouts at home. We will ensure participants are physically able to embark on this by taking their medical history, physical examination and validated questionnaire (PARQ). This program is for the benefit on the patients' long term health.
2. MR imaging to assess fat: occassionally these may pick up anomalies which require further investigation. A radiologist will screen the abdominal images and GP will be informed on anything requiring further investigation.

   No radiation is received during MR imaging.
3. Physiological studies: Patients will be asked to attend for 2 non-consecutive days before and after the exercise intervention. Regular blood samples will be required as apart of these investigations.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary, non smoking, male subjects,
* Alcohol consumption men <21 units/week,
* BMI 27-35. (Lean individuals do not suffer from NAFLD, so are not suitable for this study. Conversely, we are restricted to a maximum BMI of 35 due to the size limitations of the MR scanner.)
* A clinical diagnosis of NAFLD based upon the following criteria: i) exclusion of other causes of liver disease i.e. negative Hepatitis B and C serology, a negative auto-immune profile and normal caeruloplasmin concentrations, ii) Ultrasound appearances suggestive of a fatty, echo-bright liver with no evidence of cirrhosis (in some cases, the diagnosis will have been confirmed histologically after liver biopsy.
* Being willing to engage and motivated to follow an exercise program.

Exclusion Criteria:

* Prescription of corticosteroids, amiodarone, tamoxifen, methotrexate (drugs known to cause secondary steatohepatitis) or fibrates. Statin is Ok as long as the patients are on stable therapy for a while, if changed then the patient will be excluded.
* Alcohol consumption for men 21 units/week.
* A contraindication to exercise (such as unstable ischaemic heart disease),
* Type 2 diabetes (type 2 diabetes patients are excluded so that we are examining the involvement of insulin resistance at a reversible stage before β-cell failure has occurred).
* Patients who are on medications that will interact with GTN (glyceryl trinitrate) will be excluded from the GTN dilatation (endothelial independent NO mediated function) aspect of the study.
* Individuals who suffer from claustrophobia and have metal implants will be excluded from the MRI aspect of the study.
* Patients who smoke will also be excluded from the study.
* Total cholesterol >7

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2013-04-01 (Actual); Study Completion 2013-04-01 (Actual)

PRIMARY OUTCOMES:
Reduction in liver and muscle fat | 4 months
  Tissue triglyceride content, or steatosis, will be accurately and non-invasively quantified in vivo using localized proton magnetic resonance spectroscopy (1H MRS).

SECONDARY OUTCOMES:
Changes in liver function tests | 4 months
  Biochemial measurements of the liver enzymes will be measured pre and post intervention period
Changes in lipid profiles | 4 months
  Total cholesterol, triglyceride and high density lipoprotien concentrations in fasting state will be measured pre and post intervention period.
Changes in body weight and anthropometric measurements | 4 months
  Body weight and waist to hip ratio will be measured pre and post intervention period.
Hepatic insulin sensitivity | 4 months
  Half of the study cohort i.e. 30 individuals,15 exercise and 15 controls, will have peripheral and hepatic insulin sensitivity determined using a two-stage hyperinsulinaemic, euglycaemic clamp and use of deuterated glucose (2H2-glucose
VLDL-TG kinetics | 4 months
  The other half of the study cohort i.e. 30 individuals, 15 exercise and 15 controls, will have VLDL1 and VLDL2 TG kinetics determined using 5H2 glycerol bolus.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cuthbertson, BSc PhD MRCP, Study Director — University of Liverpool; Fariba Shojaee-Moradie, BSc PhD, Principal Investigator — University of Surrey
Locations (7):
- United Kingdom (7):
  - Royal Surrey County Hospital, Guildford, Surrey
  - University of Surrey, Guildford, Surrey
  - John Moores University, Liverpool
  - University of Liverpool, Liverpool
  - Royal Liverpool University Hospital, Liverpool
  - Liverpool University, Liverpool
  - Imperial College London, London

REFERENCES:
- [Derived] Shojaee-Moradie F, Cuthbertson DJ, Barrett M, Jackson NC, Herring R, Thomas EL, Bell J, Kemp GJ, Wright J, Umpleby AM. Exercise Training Reduces Liver Fat and Increases Rates of VLDL Clearance But Not VLDL Production in NAFLD. J Clin Endocrinol Metab. 2016 Nov;101(11):4219-4228. doi: 10.1210/jc.2016-2353. Epub 2016 Sep 1. PMID 27583475
- [Derived] Pugh CJ, Sprung VS, Jones H, Richardson P, Shojaee-Moradie F, Umpleby AM, Green DJ, Cable NT, Trenell MI, Kemp GJ, Cuthbertson DJ. Exercise-induced improvements in liver fat and endothelial function are not sustained 12 months following cessation of exercise supervision in nonalcoholic fatty liver disease. Int J Obes (Lond). 2016 Dec;40(12):1927-1930. doi: 10.1038/ijo.2016.123. Epub 2016 Jul 21. PMID 27439593